CLINICAL TRIAL: NCT02557113
Title: Creation of a Small Cavity in Vertebral Body Reduces the Rate of Cement Leakage During Vertebral Body Augmentation: A Prospective Randomized Controlled Study
Brief Title: Creation of a Small Cavity Reduces the Rate of Cement Leakage During Vertebral Body Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad ARAB MOTLAGH (Other)
Responsible Party: Sponsor-Investigator, Mohammad ARAB MOTLAGH, Dr. med., Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cavuplasty
Record Dates: First submitted 2015-09-20; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Vertebral Body Fracture
Keywords: cement leakage; cement augmentation; vertebral body fracture; vertebral cavity; vertebroplasty
MeSH Terms: interventions — Vertebroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vertebroplasty (Active Comparator): This Group Underwent the Vertebroplasty Procedure (Injection of Bone Cement into the Fractured Osteoporotic Vertebral Body)
  Interventions: Procedure: Vertebroplasty
- Cavuplasty (Experimental): This Group Underwent the Cavuplasty Procedure (Small Cavity was Created in the Vertebral Body Prior to Injection of Bone Cement)
  Interventions: Procedure: Cavuplasty

INTERVENTIONS:
Procedure: Vertebroplasty — Fractured Osteoporotic Vertebral Body is Augmented with Injection of Bone Cement
  Arms: Vertebroplasty
Procedure: Cavuplasty — Small Cavity is Created in Fractured Osteoporotic Vertebral Body Prior to Cement Injection
  Arms: Cavuplasty

SUMMARY:
Leakage of polymethylmethacrylate (PMMA) is the most common complication during vertebral body augmentation and can lead to serious patient morbidity. Any measure to reduce the rate of cement leakage is of value and makes the procedure safer.The aim of this study was to investigate the effect of the creation of a cavity on cement leakage during vertebroplasty. Investigators tested the hypothesis that the creation of a merely small and irregular cavity in vertebral body prior to cement injection would reduce cement leakage.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic vertebral body fractures of the thoracolumbar spine (T9 to L4) that were classified as A1 fractures according to Arbeitsgemeinschaft Osteosynthesis (AO) Classification

Exclusion Criteria:

* More Than 2 Vertebral Body Fractures
* Fractures of Vertebral Body Based on Malignancy
* Previous Spinal Operation
* Spinal Infection
* Spinal Deformity (scoliosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
CT-Scan evaluation | One week
  Number of Cement Extravasation in each Vertebral Body

SECONDARY OUTCOMES:
Visual Analogue Scale | 3 Months
  Scores range from 0 (no pain) to 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arab Motlagh, MD, Study Director — Department of Orthopaedic Surgery University Hospital Frankfurt